CLINICAL TRIAL: NCT03409185
Title: The Incidence of Glistenings in the 2017 Generation of Hydrophobic Acrylic Lenses Manufactured by Alcon and Abbott Medical Optics
Brief Title: The Incidence of Glistenings in the 2017 Intraocular Lenses Made by Alcon and Abbott Medical Optics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of low recruitment/enrolment due to multiple reasons, including 1) Elderly population, often with other health issues, thus not being able to commit to all of the follow-up appointments and 2) COVID-19 restrictions.
Sponsor: University of Toronto (Other)
Collaborators: Kensington Eye Institute (Other)
Responsible Party: Principal Investigator, Yaping Jin, Associate Professor in Ophthalmic Epidemiology, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 108162330RR0001
Record Dates: First submitted 2017-12-18; First posted 2018-01-24 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Cataracts; Visual Acuity Reduced Transiently; Loss of Visual Contrast Sensitivity; Functional Visual Loss
Keywords: Cataract surgery; Intraocular lens; Glistenings
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Alcon lens group (Experimental): Alcon 1 piece SA60AT lens
  Interventions: Device: Alcon 1 piece SA60AT lens
- AMO lens group (Active Comparator): AMO 1 piece Sensar AABOO lens
  Interventions: Device: AMO 1-piece AABOO lens

INTERVENTIONS:
Device: Alcon 1 piece SA60AT lens — Optic Diameter: 6.0 mm, Overall length: 13.0 mm, Material: Ultraviolet-absorbing Acrylate/Methacrylate Copolymer
  Arms: Alcon lens group
Device: AMO 1-piece AABOO lens — Optic Diameter: 6.0 mm, Overall length: 13.0 mm, Material: Ultraviolet-blocking hydrophobic acrylic
  Arms: AMO lens group

SUMMARY:
The purpose of this study is to seek academic/non-industry research funding support to independently investigate the incidence and density of lens glistenings in cataract patients who are implanted with the latest generations of intraocular lenses (IOL) manufactured by Alcon and AMO Medical Optics.

DETAILED DESCRIPTION:
Glistenings are tiny, clear sparkling, fluid-filled microvacuoles that form within a lens after it has been placed in the eye. Glistenings are seen in all lenses but certain lenses develop a higher number of glistenings than others. The effect of glistenings on patients' visual functioning is largely unknown.

The occurrence of glistenings is in part related to the manufacturing technique. In 2013, manufacturers have claimed that recent improvements in manufacturing process have reduced the occurrence of glistenings. There is a lack of independent evaluation of this claim. We would like to assess independently: 1) How frequently do glistenings occur in patients implanted with the 2015 generation lenses? 2) Is there a difference in glistening occurrence between lenses manufactured by Alcon and Abbott Medical Optics (AMO) - the two largest companies in eye care products?

Two-hundred and seventy-six patients will be randomly assigned to receive Alcon or AMO lenses for their cataract surgery at the Kensington Eye Institute (KEI). After surgery, patients will be instructed to return for follow-up visits at 1 month, 6 months, 12 months and 18 months to assess for the occurrence of glistenings. If glistenings are observed at an earlier follow-up visit (e.g., the 6 month visit), patients will still be instructed to come for future visits so that changes in the glistenings over time can be observed.

Project Time-line:

Months 1-8: Participants recruiting, surgical operations, follow-up visits. Months 9-24: follow-up visits, data entry, cleaning and analysis, early results presentation, manuscript preparation and final report.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting 5 surgeons for cataract surgery in the surgeon's primary offices
* Patients aged 18 years or older
* Patients who signed the consent form

Exclusion Criteria:

* Individuals who cannot understand English in either written or verbal form and do not have language assistance available (e.g. from family members, friends)
* Patients with co-existing condition of corneal disease
* Patients with co-existing condition of uveitis
* Patients with co-existing condition of optic nerve disease
* Patients with co-existing condition of macular disease
* Patients with co-existing condition of diabetes
* Patients with co-existing condition of severe glaucoma (i.e. C/D ratio >=0.9 AND the patient is on glaucoma treatment)
* Patients with prior refractive surgery
* Patients with complications of cataract surgery occurred during or after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence and density (severity) of glistenings at 18-month follow-up visit | 18-month follow-up
  To determine if glistenings develop, eyes are dilated and examined. Photographs of the IOLs will be taken with a slit lamp camera for documentation. These photographs will then be assessed for glistenings in two ways: first by trained ophthalmology staff, and second using the ImageJ software
  Glistenings will be counted and graded on a scale of 0 to 5+ as following:
  0. No glistening
  1. Less than 10 glistenings
  2. 10 to 25 glistenings
  3. 25 to 50 glistenings
  4. 50 to 100 glistenings
  5. Greater than 100 glistenings

SECONDARY OUTCOMES:
Visual acuity in eyes with glistenings at 18-month follow-up visit | 18 month follow-up
  Best corrected visual acuity: acuteness/clearness of vision. This will be tested with the ETDRS (early treatment diabetic retinopathy study) chart.
Contrast sensitivity in eyes with glistenings at 18-month follow-up visit | 18 month follow-up
  Contrast sensitivity: the ability of the visual system to distinguish between an object and its background. This will be tested with the Vector Vision CSV-1000HGT.
Glare disability in eyes with glistenings at 18-month follow-up visit | 18 month follow-up
  Glare disability: the difficulty seeing in the presence of very bright light such as night-time lighting or sunshine. This will be tested using the Brightness Acuity Tester (BAT).
Visual acuity in eyes with glistenings at 12-month follow-up visit | 12-month follow-up
  Best corrected visual acuity: acuteness/clearness of vision. This will be tested with the ETDRS (early treatment diabetic retinopathy study) chart
Contrast sensitivity and glare disability in eyes with glistenings at 12-month follow-up visit | 12-month follow-up
  Contrast sensitivity: the ability of the visual system to distinguish between an object and its background. This will be tested with the Vector Vision CSV-1000HGT.
Glare disability in eyes with glistenings at 12-month follow-up visit | 12-month follow-up
  Glare disability: the difficulty seeing in the presence of very bright light such as night-time lighting or sunshine. This will be tested using the Brightness Acuity Tester (BAT).
Visual acuity in eyes with glistenings at 6-month follow-up visit | 6-month follow-up
  Best corrected visual acuity: acuteness/clearness of vision. This will be tested with the ETDRS (early treatment diabetic retinopathy study) chart.
Contrast sensitivity in eyes with glistenings at 6-month follow-up visit | 6-month follow-up
  Contrast sensitivity: the ability of the visual system to distinguish between an object and its background. This will be tested with the Vector Vision CSV-1000HGT.
Glare disability in eyes with glistenings at 6-month follow-up visit | 6-month follow-up
  Glare disability: the difficulty seeing in the presence of very bright light such as night-time lighting or sunshine. This will be tested using the Brightness Acuity Tester (BAT).
Incidence of glistenings at 12-month follow-up visit | 12-month follow-up
  To determine if glistenings develop, eyes are dilated and examined. Photographs of the IOLs will be taken with a slit lamp camera for documentation. These photographs will then be assessed for glistenings in two ways: first by trained ophthalmology staff, and second using the ImageJ software
  Glistenings will be counted and graded on a scale of 0 to 5+ as following:
  0. No glistening
  1. Less than 10 glistenings
  2. 10 to 25 glistenings
  3. 25 to 50 glistenings
  4. 50 to 100 glistenings
  5. Greater than 100 glistenings
Incidence of glistenings at 6-month follow-up visit | 6-month follow-up
  To determine if glistenings develop, eyes are dilated and examined. Photographs of the IOLs will be taken with a slit lamp camera for documentation. These photographs will then be assessed for glistenings in two ways: first by trained ophthalmology staff, and second using the ImageJ software
  Glistenings will be counted and graded on a scale of 0 to 5+ as following:
  0. No glistening
  1. Less than 10 glistenings
  2. 10 to 25 glistenings
  3. 25 to 50 glistenings
  4. 50 to 100 glistenings
  5. Greater than 100 glistenings

CONTACTS AND LOCATIONS:
Overall Officials: Sherif El-Defrawy, MD, FRCSC, Principal Investigator — University of Toronto; Yaping Jin, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Kensington Eye Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided